CLINICAL TRIAL: NCT04947592
Title: Outcome of SD-OCT Guided Oral Anti-fungal Treatment of Fungal Chorioretinitis
Brief Title: SD-OCT Guided Treatment of Fungal Chorioretinitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Associate Professor, Benha University
Other Study IDs: Hamaky13
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Fungal Retinitis
Keywords: fungal; chorioretinitis; OCT
MeSH Terms: conditions — Chorioretinitis | interventions — Fluconazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fluconazole 150 mg — fluconazole 150 MG once daily for 14 days

SUMMARY:
Fungal Chorioretinitis is a vision threatening condition.The investigators evaluate the efficacy of SD-OCT role in the treatment

DETAILED DESCRIPTION:
Baseline ,and postoperative 1 ,6 and 12 months full ophthalmic examination and SD-OCT was done.Procedure included oral fluconazole treatment 1 tablet once for 14 days

ELIGIBILITY:
Inclusion Criteria:

- fungal chorioretinitis

Exclusion Criteria:

* vitritis
* other macular lesion
* macular scar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 18 years old patient with fungal chorioretinitis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 6 months
  Change in BCVA in LOG MARS(logarithm minimum angle of resolution

SECONDARY OUTCOMES:
optical coherence tomography (OCT) foveal thickness | 6 months
  change in foveal thickness measured in micrometer

CONTACTS AND LOCATIONS:
Overall Officials: TAREK ELHAMAKY, Principal Investigator — Benha University
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates